CLINICAL TRIAL: NCT04244539
Title: Efficacy of High-intensity Laser in Jaccoud's Arthropathy in Systemic Lupus Erythematosus: a Prospective Randomized Controlled Trial
Brief Title: Efficacy of High-intensity Laser in Jaccoud's Arthropathy in Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Collaborators: Cairo University (Other); Nabil Mahmoud Abdel-Aal (Unknown)
Responsible Party: Principal Investigator, Hadaya Mosaad, lecturer, Jouf University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002616
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Musculoskeletal Diseases; Skin Diseases
MeSH Terms: conditions — Musculoskeletal Diseases; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Patients in the study group received pulsed Nd: YAG laser treatment, produced by a HIRO 3 device (ASA Laser, Arcugnano, Italy). The apparatus provided pulsed emission (1064 nm), very high peak power (3 kW), a high level of fluency (energy density; 360-1780 mJ/cm2), a short duration (120-150 μs), a mean power of 10.5 W, a low frequency (10-40 Hz), a duty cycle of about 0.1%, a probe diameter of 0.5 cm, and a spot size of 0.2 cm2 [9].
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): a received routine physical therapy program, in addition to HILT. Patients in the study group received pulsed Nd: YAG laser treatment, produced by a HIRO 3 device (ASA Laser, Arcugnano, Italy). The apparatus provided pulsed emission (1064 nm), very high peak power (3 kW), a high level of fluency (energy density; 360-1780 mJ/cm2),
  Interventions: Device: high-intensity laser Device.
- Control group (Active Comparator): The control group received traditional physical therapy program in the form of strengthening exercise, stretching , and range of motion exercise.for the affected digits and wrists. for one hour, three sessions per week for 8 weeks.
  Interventions: Device: high-intensity laser Device.

INTERVENTIONS:
Device: high-intensity laser Device. — Twenty four treatment sessions with pulsed Nd: YAG laser were applied to the subjects of the study group, three sessions per week, over 8 weeks in succession via HIRO® 3.0 device (ASAlaser, Arcugnano, Vicenza, Italy). The device gives pulsed emission (λ = 1064 nm), maximum power (3000 W), fluency range (360-1780 mJ/cm2), pulse duration (≤ 100 μs), frequency range (10-40 Hz), maximum energy per pulse (350 mJ), mean power (10.5 W), and power cycle of ~0.1%.

SUMMARY:
A randomized, controlled study with the pretest-posttest design was performed; 50 patients who were suffered from jaccoud's arthropathy and aged 30-50 years. Patients were randomly assigned into two groups: Group 1 (study group): received HILT, in addition to the routine physical therapy program. Group 2 (control group): received routine physical therapy program. All treatment interventions were applied at a frequency of three sessions per week for 8 weeks. The participants were recruited from the air forces hospital at the period from December 2018 and October 2019.

DETAILED DESCRIPTION:
A sample of 55 female patients was recruited from the Kasr El-Ani hospital outpatient clinic to be treated in the outpatient clinic, Air forces hospital, Cairo. at the period from December 2018 and July 2019 with 50 of them completing the study. They were enrolled and assessed for their eligibility to participate in the study. The patients were randomly classified into 2 groups of equal number. Group 1 (Study group): received HILT, in addition to the routine physical therapy program. Group 2 (Control group): received routine physical therapy program. The patient's age ranged from 30 to 50 years. Elapsed time since the beginning of the disease was less than 1 year. All patients received the same medication. Patients were excluded if they had one or more of the following: positive rheumatic factor, circulatory disorders, neurological disease, diabetes, pregnant woman, communication problems or skin diseases.

The participants were informed in details about the nature, purpose, and benefits of the study, they had complete right to refuse or withdraw from the study at any time, and the confidentiality of any obtained information.

Interventions Patients indiscriminately assigned to study group (Group- 1):- 25 female Patients had been dealt with a received routine physical therapy program, in addition to HILT. Patients in the study group received pulsed Nd: YAG laser treatment, produced by a HIRO 3 device (ASA Laser, Arcugnano, Italy). The apparatus provided pulsed emission (1064 nm), very high peak power (3 kW), a high level of fluency (energy density; 360-1780 mJ/cm2), a short duration (120-150 μs), a mean power of 10.5 W, a low frequency (10-40 Hz), a duty cycle of about 0.1%, a probe diameter of 0.5 cm, and a spot size of 0.2 cm2 [9]. Twenty four treatment sessions with pulsed Nd: YAG laser were applied to the subjects of the study group, three sessions per week, over 8 weeks in succession via HIRO® 3.0 device (ASAlaser, Arcugnano, Vicenza, Italy). The device gives pulsed emission (λ = 1064 nm), maximum power (3000 W), fluency range (360-1780 mJ/cm2), pulse duration (≤ 100 μs), frequency range (10-40 Hz), maximum energy per pulse (350 mJ), mean power (10.5 W), and power cycle of ~0.1%. The device is equipped with a standard handpiece endowed with a fixed spacer and has a diameter of 0.5 cm and a spot size of 0.2 cm2. A pair of protective eye goggles were provided for the both the participant and the therapist. The participants were treated while assuming a sitting position, with their hand rested at the table. Every laser application comprised three phases: phase 1, where a fast scanning was applied transversely and longitudinally around the wrist and hand with three respective fluencies set at 510, 610, and 710 mJ/cm2 for a total of 300 J; phase 2, where a total of 10 fixed points around metacarpophalangeal joint and wrist joint were irradiated, in this phase, each point was radiated for 15 s, using a fluency of 710 mJ/cm2, 150 J/point, and a total of 150 J; and phase 3, where a scanning like that in phase 1 was applied, but at a much slower rate with a total energy of 300 J. The scanning energy density was 10 J/cm2 and the average irradiated area was 60 cm2. The control group (Group 2): 25 female Patients, in Group-B had been dealt with routine physical therapy program for 8 weeks, 3 sessions /week. Both groups received 24 sessions of treatment, 3 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranged from 30 to 50 years.
* Elapsed time since the beginning of the disease was less than 1 year.
* All patients received the same medication

Exclusion Criteria:

* Patients were excluded if they had one or more of the following:
* Positive rheumatic factor,
* Circulatory disorders,
* Neurological disease,
* Diabetes,
* Pregnant woman,
* Communication problems
* Skin diseases.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | after 8 weeks of intervention.
  Handheld Jamar dynamometer device 12-0600 was used to measure handgrip strength. The readout of dynamometer dial is represented in pounds and in kilograms. It is graded from zero to two hundred pounds and from zero to ninety kilograms [14]. Grip measurement was performed with the elbow at about 90° according to the American Society of Hand Therapists (ASHT) recommendations .The patients were instructed to assume the sitting position while the affected limb was placed in shoulder adduction and internal rotation, elbow flexion, forearm in mid-position and wrist in the neutral position. The patients were instructed to squeeze the dynamometer as much as possible. Three consecutive measurements were performed with a 2 minutes inter-measurement interval.

SECONDARY OUTCOMES:
Joint counts for tenderness and swelling | after 8 weeks of intervention
  the sum of the number of affected joints
Pain Intensity: visual analogue scale (VAS) | after 8 weeks of treatment.
  A visual analogue scale (VAS) was used for the assessment of joint pain [17]. It is an ordinal scale, using a 100-mm line divided into 10 equal sections, with 0 representing "no pain" and 10 representing "unbearable pain." Each participant was asked to indicate on the scale the level of pain in the hand and wrist joint at the baseline and post-treatment after the end of sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Abdel-Aal, Assist.prof., Study Director — Cairo University, Faculty of physical Therapy.
Locations (1):
- Faculty of physical therapy, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and informed Consent form will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: we will share results after 6 months of publication.